CLINICAL TRIAL: NCT07163221
Title: At-home Ultrasound Localized Therapy for Rheumatoid Arthritis Study [At-home ULTRA Study]
Acronym: At-home ULTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SecondWave Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00087265
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: RA; SecondWave Systems; SecondWave; Rheumatoid Arthritis; Neuromodulation; Ultrasound; Splenic Ultrasound; Spleen; Spleen stimulation; Ultrasound Stimulation; Immunomodulation; spleen stimulating device; drug refractory; noninvasive; non-invasive
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: A 2-stage, randomized, double-blind, sham-controlled, multicenter study. Participants will be randomized into three groups, where one group is the standard of care control and the other two groups are standard of care plus differing stimulation settings of the SecondWave MINI therapy. Participants assigned to the treatment group will receive active stimulation for 20 min once per day, and those assigned to the control group will receive sham-stimulation for 20 min once per day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, joint evaluators and outcome assessors will be blinded. Blinding of subjects will be assessed at Week 12.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Control (Sham Comparator): Non-active Sham Stimulation
  Interventions: Device: Sham ultrasound stimulation (control); Drug: Conventional Synthetic DMARD
- Treatment Setting 1 (Experimental): Subjects will receive daily noninvasive ultrasound stimulation of the spleen using Ultrasound Treatment Setting 1 for 20 minutes once per day
  Interventions: Device: Non-invasive ultrasound stimulation of the spleen - Treatment Setting 1; Drug: Conventional Synthetic DMARD
- Treatment Setting 2 (Experimental): Subjects will receive daily noninvasive ultrasound stimulation of the spleen using Ultrasound Treatment Setting 2 for 20 minutes once per day
  Interventions: Device: Non-invasive ultrasound stimulation of the spleen - Treatment Setting 2; Drug: Conventional Synthetic DMARD

INTERVENTIONS:
Device: Non-invasive ultrasound stimulation of the spleen - Treatment Setting 1 — Subjects will receive daily noninvasive ultrasound stimulation of the spleen using Ultrasound Treatment Setting 1 for 20 minutes once per day
  Arms: Treatment Setting 1
Device: Non-invasive ultrasound stimulation of the spleen - Treatment Setting 2 — Subjects will receive daily noninvasive ultrasound stimulation of the spleen using Ultrasound Treatment Setting 2 for 20 minutes once per day
  Arms: Treatment Setting 2
Device: Sham ultrasound stimulation (control) — Sham ultrasound stimulation for 20 minutes once per day
  Arms: Control
Drug: Conventional Synthetic DMARD — All subjects will take at least one type of conventional synthetic DMARD at the same stable dose for at least 8 weeks prior to the treatment period and continuing through study close out

SUMMARY:
The At-Home ULTRA Study will evaluate performance of the MINI system as indicated for the treatment of adults with active, moderate to severe rheumatoid arthritis who are inadequate responders or are intolerant to conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs), biologic DMARDs (bDMARDs), or targeted synthetic DMARDs (tsDMARDs). The non-invasive study device delivers ultrasound stimulation to the spleen to reduce inflammation. The study will enroll at least 60 participants at up to 8 sites. There will be three arms consisting of two active stimulation groups (treatment) and one non-active stimulation group (sham-control). After completing the double-blinded primary endpoint assessment period at Week 12, there will be a one-way crossover of control participants to active stimulation and an additional 12 week follow-up with all participants to evaluate long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18 and above
2. Active moderate to severe seropositive RA
3. At least 6 total tender and/or swollen joints counted on a 28 joint assessment during screening and at Week 0 (a joint that is both tender and swollen will be counted as "2")
4. Demonstrated an inadequate response to, or loss of response to standard csDMARD treatment (e.g., methotrexate) or up to three total bDMARDs and tsDMARDs
5. Receiving stable background treatment with a csDMARD prior to start of the treatment period at Week 0. Methotrexate (if chosen as background treatment) must be maintained at a stable dose for at least 4 weeks prior to Week 0, while all other csDMARDs (if chosen as background treatment) must be maintained at a stable dose for at least 8 weeks prior to Week 0. Participants must be willing to maintain their background medication regimen throughout the 28-week study period.
6. For participants that have previously undergone treatment with bDMARDs or tsDMARDs therapy, those treatments must be discontinued at least 4 weeks prior to start of the treatment period at Week 0 and may not be resumed until after the Week 24 Closeout Visit
7. For participants that have previously undergone treatment with Golimumab or Infliximab, those treatments must be discontinued at least 8 weeks prior to start of the treatment period at Week 0 and may not be resumed until after the Week 24 Closeout Visit
8. Participants may receive up to 10 mg of daily prednisone as part of their background treatment but must have maintained a stable dose for a minimum of 6 weeks prior to start of the treatment period at Week 0, and must be willing to maintain the stable dose until after the Week 24 Closeout Visit
9. Torso circumference at the belly button and sternum level must both be in the range of 25 to 50 inches
10. Participants with an immunomodulation device must be willing and able to turn the device off at least 4 weeks prior to start of the treatment period at Week 0 and may not be resumed until after the Week 24 Closeout Visit
11. Participants must be willing not to initiate any new treatments with expected immune modulating effects during the study period, and any existing immune modulating treatments must be stabilized by Week 0
12. Participants must be willing and able to follow the medication rules described in the study's IRB-approved Medication Guide

Exclusion Criteria:

1. Active bacterial or viral infection
2. Pregnant women or those trying to become pregnant
3. Receiving active chemotherapy or immunotherapy to treat malignancy within 30 days prior to enrollment
4. Having received more than a total of three bDMARDs and tsDMARDs
5. Having received Rituximab monoclonal antibody medication
6. Presence of an implanted device or other solid object in the vicinity of the spleen that can interfere with or absorb the ultrasound beam
7. History of asplenia
8. History of splenomegaly
9. History of ascites
10. Recent abdominal surgery
11. Currently participating in an investigational drug or device study
12. Open wound/sores that would make performing study procedures too difficult
13. Inability to perform minimal daily self-cares associated with feeding or dressing, such as lifting a cup of water to the mouth or putting on clothing.
14. Refusal or inability to regularly attend the scheduled on-site visits and at-home visits, or perform the remote video observation sessions
15. Cannot speak English
16. Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in DAS28-CRP score from baseline to 12 weeks, compared between Arm 1 and Arm 3 (sham control) | 12 weeks
  A decrease in Disease Activity Score indicates an improved outcome
Change in DAS28-CRP score from baseline to 12 weeks , compared between Arm 2 and Arm 3 (sham control) | 12 weeks
  A decrease in Disease Activity Score indicates an improved outcome

OTHER OUTCOMES:
Comparison of responder rate between Arm1 or Arm 2 versus Arm 3 for the ACR20 | 12 and 24 weeks
  ACR20, the American College of Rheumatology (ACR) 20 response is defined as 20% improvement in tender and swollen joint counts and 20% improvement in 3 of the 5 remaining ACR core set measures: patient and physician global assessments, pain, disability, and an acute-phase reactant
Comparison of responder rate between Arm1 or Arm 2 versus Arm 3 for the ACR50 | 12 and 24 weeks
  ACR50, the American College of Rheumatology (ACR) 50 response is defined as 50% improvement in tender and swollen joint counts and 50% improvement in 3 of the 5 remaining ACR core set measures: patient and physician global assessments, pain, disability, and an acute-phase reactant
Comparison of responder rate between Arm1 or Arm 2 versus Arm 3 for the ACR70 | 12 and 24 weeks
  ACR70, the American College of Rheumatology (ACR) 70 response is defined as 70% improvement in tender and swollen joint counts and 70% improvement in 3 of the 5 remaining ACR core set measures: patient and physician global assessments, pain, disability, and an acute-phase reactant
Good EULAR response | 12 and 24 weeks
  European Alliance of Associations for Rheumatology (EULAR) "good" response corresponding to clinical improvement in patients with rheumatoid arthritis (RA) and is defined by a DAS28-CRP of ≤3.2 and a DAS28-CRP decrease of more than 1.2 from the baseline score
Moderate EULAR response | 12 and 24 weeks
  European Alliance of Associations for Rheumatology (EULAR) "moderate" response corresponding to clinical improvement in rheumatoid arthritis (RA) and is defined as either a decrease in DAS28-CRP of >0.6 to ≤1.2 while maintaining a DAS28 score of ≤5.1, OR a decrease of >1.2 in DAS28-CRP but with a current score >3.2
Satisfaction response | 12 and 24 weeks
  Questions to assess benefit, acceptance and usability of the treatment
Change in HAQ-DI | 12 and 24 weeks
  The Health Assessment Questionnaire Disability Index (HAQ-DI) is made up of 8 domains of daily activity. A decrease in score indicates improved physical function
Change in DAS28-CRP score from baseline to 24 weeks, compared between Arm 1 and Arm 3 (sham control) | 24 weeks
  A decrease in Disease Activity Score indicates an improved outcome
Change in DAS28-CRP score from baseline to 24 weeks, compared between Arm 2 and Arm 3 (sham control) | 24 weeks
  A decrease in Disease Activity Score indicates an improved outcome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zachs, Study Director — SecondWave Systems Inc.
Locations (5):
- United States (5):
  - Arizona Arthritis and Rheumatology Associates P.C., Glendale, Arizona
  - Medvin Clinical Research, Covina, California
  - Southland Arthritis & Osteoporosis Medical Center, Temecula, California
  - University of Colorado, Aurora, Colorado
  - University of Minnesota Medical School, Division of Rheumatic and Autoimmune Diseases, Minneapolis, Minnesota